CLINICAL TRIAL: NCT03958396
Title: The Pharmacokinetic and Pharmacodynamics Profiles of Remifentanil in Children With Obstructive Sleep Apnea.
Brief Title: Remifentanil in Children With Obstructive Sleep Apnea
Acronym: ROSA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201504056
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Parallel group study comparing patients with obstructive sleep apnea undergoing tonsillectomy or tonsillectomy and adenoidectomy to controls with no history of obstructive sleep apnea undergoing general anesthesia for any procedure. The study will be conducted in the patient's preoperative holding area room. Two intravenous catheters will be placed, one for a remifentanil infusion and one for blood draws to measure the blood concentration of remifentanil. Patients will have standard ASA monitors placed with vital signs monitored on a portable monitor, and a remifentanil infusion will be started. Blood draws will be taken at seven time points: zero, one, two, four, six, ten and fifteen minutes. Concomitantly, recordings of end tidal CO2, respiratory rate, and pupil diameter will be made at the seven time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- OSA Group (Active Comparator): a) Children 8-14 years old, b) ASA physical status 1or 2, c) undergoing tonsillectomy or tonsillectomy and adenoidectomy for known obstructive sleep apnea
  Interventions: Drug: Remifentanil Infusion
- Control (non-OSA) Group (Active Comparator): a) Children 8-14 years old, b) ASA physical status 1or 2, c) no known obstructive sleep apnea presenting for any procedure requiring general anesthetic
  Interventions: Drug: Remifentanil Infusion

INTERVENTIONS:
Drug: Remifentanil Infusion — 15 minute remifentanil Infusion of either 0.05, 0.1, 0.15 or 0.2 mcg/kg/min

SUMMARY:
This investigation tested the hypothesis that children with obstructive sleep apnea have an increased pharmacodynamic sensitivity to the miotic and respiratory depressant effects of the prototypic μ-opioid agonist remifentanil.

ELIGIBILITY:
OSA Group:

Inclusion Criteria:

* 8-14 years old
* ASA physical status 1 or 2
* undergoing tonsillectomy or tonsillectomy and adenoidectomy for known obstructive sleep apnea

Exclusion Criteria:

* Inability to cooperate with study requirements (IV placement, sitting quietly, wearing goggles, etc.)

Control (Non-OSA) Group:

Inclusion Criteria:

* 8-14 years old
* ASA physical status 1 or 2
* no known obstructive sleep apnea presenting for any procedure requiring general anesthtic

Exclusion Criteria:

* Inability to cooperate with study requirements (IV placement, sitting quietly, wearing goggles, etc.)

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Change in end-expired carbon dioxide from baseline over time - OSA Group | Approximately 1 hour before surgery - Measurements taken at 0, 1, 2, 4, 6, 10 & 15 minutes following remefentanil infusion
  End-expired carbon dioxide monitoring using bedside monitoring
Change in end-expired carbon dioxide from baseline over time - Control (non-OSA) Group | Approximately 1 hour before surgery - Measurements taken at 0, 1, 2, 4, 6, 10 & 15 minutes following remefentanil infusion
  End-expired carbon dioxide monitoring using bedside monitoring
Change in respiratory rate from baseline over time - OSA Group | Approximately 1 hour before surgery - Measurements taken at 0, 1, 2, 4, 6, 10 & 15 minutes following remefentanil infusion
  Respiratory monitoring was performed using nasal cannula
Change in respiratory rate from baseline over time - Control (non-OSA) Group | Approximately 1 hour before surgery - Measurements taken at 0, 1, 2, 4, 6, 10 & 15 minutes following remefentanil infusion
  Respiratory monitoring was performed using nasal cannula
Change in pupil diameter from baseline over time - OSA Group | Approximately 1 hour before surgery - Measured continuously and averaged into 10-s bins following remefentanil infusion
  Dark adapted infrared pupillometry performed using binocular infrared pupilometer mounted in light occlusive goggles sampling at 100 Hz.
Change in pupil diameter from baseline over time - Control (non-OSA) Group | Approximately 1 hour before surgery - Measured continuously and averaged into 10-s bins following remefentanil infusion
  Dark adapted infrared pupillometry performed using binocular infrared pupilometer mounted in light occlusive goggles sampling at 100 Hz.
Remifentanil plasma concentration - OSA Group | Approximately 1 hour before surgery - Blood draws at 0, 1, 2, 4, 6, 10 & 15 minutes following remefentanil infusion
  3ml blood draw
Remifentanil plasma concentration - Contro (non-OSA) Group | Approximately 1 hour before surgery - Blood draws at 0, 1, 2, 4, 6, 10 & 15 minutes following remefentanil infusion
  3ml blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Anshuman Sharma, MD, Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Result] Brown KA. Outcome, risk, and error and the child with obstructive sleep apnea. Paediatr Anaesth. 2011 Jul;21(7):771-80. doi: 10.1111/j.1460-9592.2011.03597.x. Epub 2011 May 3. PMID 21539679
- [Result] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Ward SD, Sheldon SH, Shiffman RN, Lehmann C, Spruyt K; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):e714-55. doi: 10.1542/peds.2012-1672. Epub 2012 Aug 27. PMID 22926176
- [Result] Bhattacharyya N, Lin HW. Changes and consistencies in the epidemiology of pediatric adenotonsillar surgery, 1996-2006. Otolaryngol Head Neck Surg. 2010 Nov;143(5):680-4. doi: 10.1016/j.otohns.2010.06.918. PMID 20974339